CLINICAL TRIAL: NCT02899468
Title: Evaluation of a Novel Integrative and Intensive Virtual Rehabilitation Program for Service Members Post TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Bright Cloud International Corp (Industry); Walter Reed National Military Medical Center (U.S. Federal Agency); Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 412759
Record Dates: First submitted 2016-08-24; First posted 2016-09-14 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Traumatic Brain Injury
Keywords: TBI; Virtual Reality
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Treatment Group (Experimental): Active treatment will consist of the BrightBrainer Virtual Reality (BBVR) Rehabilitation System therapy intervention (3 sessions per week x 6 weeks). Standard validated outcome measures which assess various domains of function, will be obtained at baseline and then at 3 and 6 weeks for those randomized to the Active Treatment group.
  Interventions: Device: BrightBrainer Virtual Reality (BBVR) Rehabilitation System
- Wait-List Control Group (Other): Subjects randomized to the Wait-List Control (WLC) group will wait 3 weeks before beginning the Active Treatment program intervention (3 sessions per week x 6 weeks) using the BrightBrainer Virtual Reality (BBVR) Rehabilitation System. For those randomized to the WLC group, outcome measures will be assessed at baseline, completion of waiting period (3 weeks), then at 3 and 6 weeks after initiating active treatment.
  Interventions: Device: BrightBrainer Virtual Reality (BBVR) Rehabilitation System

INTERVENTIONS:
Device: BrightBrainer Virtual Reality (BBVR) Rehabilitation System — During the active treatment stage (3 sessions per week x 6 weeks), each BBVR therapy session will consist of a series of custom games targeting one or several cognitive domains of executive function, attention, short-term memory, working memory and language comprehension. In addition, the BBVR device incorporates uni- and bi-manual activities by having the subject manipulate hand-held devices, which are programmed to measure in real time the subject's 3D hand movement and index flexion/extension. Therefore, in addition to completing the cognitive tasks, subjects must manipulate virtual hands through a hand-held interface to also enhance visual-motor perception, hand-eye coordination, and upper limb function. In addition, wrist weights can be added to increase upper limb strength training.

SUMMARY:
The purpose of the study is to evaluate the feasibility and effectiveness of a novel virtual reality (VR) therapeutic rehabilitative device (BrightBrainerTM) to treat patients with traumatic brain injury (TBI). These patients, service members with TBI, can be both with and without upper limb dysfunction and use uni- and bimanual virtual reality (VR) exercises to improve cognitive and motor function, as well as mood.

DETAILED DESCRIPTION:
Bright Cloud International Corp created BrightBrainer, a computerized virtual reality system that provides a combination of cognitive as well as motor skill training in an engaging and repetitive manner [1]. This project objective is to assess the feasibility and clinical benefit of utilizing the BBVR to augment the rehabilitation of service members with TBI. The BrightBrainerTM Virtual Reality (BBVR) Rehabilitation System is unique because it is designed to provide integrative, customized, intensive and self-guided therapy that simultaneously addresses the cognitive, emotive and motor deficits. Early evidence suggests that it has been effective for patients with cognitive deficits as the result of cerebrovascular accident or dementia, but has not yet been evaluated in a therapeutic intervention for patients with TBI. In addition to assessing the system's effect on patient's symptoms, we will also evaluate the feasibility of utilizing this system in a military environment by obtaining feedback from the patients and therapists, regarding system acceptance, reliability and ease of use.

ELIGIBILITY:
Inclusion Criteria:

* Male or female military health care beneficiaries 18-67 years of age;
* Presence of TBI (based on standard Veterans Affairs (VA)/ Department of Defense (DoD) criteria);
* With or without upper extremity dysfunction. Upper extremity dysfunction includes but is not limited to decreased coordination, increased tone, decreased strength, and decreased sensation;
* Ability to follow study instructions and likely to complete all required visits for the study;
* Ability to understand spoken and written English;
* At least 6 weeks post TBI.

Exclusion Criteria:

* Age less than 18 or greater than 67;
* Blind or otherwise visually impaired to the extent that lack of sight inhibits utilizing the system;
* Deafness;
* Inability to understand or comprehend consenting to the study;
* Active psychosis, suicidal or homicidal ideations or frequent violent episodes;
* Currently enrolled in active substance abuse treatment
* Inability to even minimally operate BBVR controllers.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-01; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Feasibility of integration of two side-by-side BrightBrainer Virtual Reality (BBVR) Rehabilitation Systems into the clinical rehabilitation practice at Walter Reed National Military Medical Center. | At the midpoint (3 weeks)
  Clinician Feedback Questionnaire: In order to determine technology feasibility and technology acceptance by the healthcare provider, we will use a subjective evaluation rating questionnaire. The rating will be similar to that used in the subjects' questionnaire, however, questions will differ.
Feasibility of integration of two side-by-side BBVR systems into the clinical rehabilitation practice at Walter Reed National Military Medical Center. | At the endpoint (6 weeks)
  Clinician Feedback Questionnaire: In order to determine technology feasibility and technology acceptance by the healthcare provider, we will use a subjective evaluation rating questionnaire. The rating will be similar to that used in the subjects' questionnaire, however, questions will differ.

SECONDARY OUTCOMES:
Subject and clinician acceptance of the BBVR system (ease of use, ease of set up and monitoring, ease of data report production, ease of monitoring two subjects simultaneously) | At the midpoint (3 weeks) of the active treatment for every participant.
  Technology Acceptance Questionnaire. To determine technology acceptance by subjects we will use a subjective evaluation rating questionnaire. The rating will be done using a 7-point Likert scale.
Subject and clinician acceptance of the BBVR system (ease of use, ease of set up and monitoring, ease of data report production, ease of monitoring two subjects simultaneously) | At the endpoint (6 weeks) of the active treatment for every participant.
  Technology Acceptance Questionnaire. To determine technology acceptance by subjects we will use a subjective evaluation rating questionnaire. The rating will be done using a 7-point Likert scale.
Participant cognitive performance | Change in performance from baseline to completion of the wait-list (for the wait-list control group only), and end point (6 weeks) of active treatment.
  Neurocognitive Assessment. The Automated Neuropsychological Assessment Metrics (ANAM) is a library of 22 computer-based assessments that are sensitive to cognitive change in attention, concentration, reaction time, memory, processing speed, and decision-making.
  Performance will also be gauged by recording subjects' performance on the BBVR.
Participant motor function (range of motion, strength, and coordination) - Fugl-Meyer Assessment | Change in functional performance from baseline to completion of the wait-list (for the wait-list control group only), and end point (6 weeks) of active treatment.
  Subjects will complete the Fugl-Meyer Assessment that measures range of motion, strength and coordination. Strength will be measured using isometric or isotonic measures of shoulder abduction, shoulder flexion, and shoulder rotation.
Participant motor function - Jebsen Hand Function Test | Change in functional performance from baseline to completion of the wait-list (for the wait-list control group only), and end point (6 weeks) of active treatment.
  Subjects will be administered the Jebsen Hand Function Test (JHFT). The JHFT is a clinically validated hand function test developed by Jebsen, Taylor, Treischmann, Trotter, and Howard in 1969. It is a standardized evaluative measure of functional hand motor skills, and consists of 7 timed tasks - that measure a) fine motor skills, b) weighted functional tasks, and c) non-weighted functional tasks.
Participant motor function - Box and Blocks Test | Change in functional performance from baseline to completion of the wait-list (for the wait-list control group only), and end point (6 weeks) of active treatment.
  Subjects will also be administered the Box and Blocks Test (BBT). The BBT measures gross manual dexterity and will be conducted bilaterally for the purpose of this study. The assessment consists of a wooden box divided into two compartments by a partition and 150 blocks. Subjects will be asked to move, one by one, blocks from one compartment of a box to another. For the purpose of this study, subjects will be presented with two boxes and asked to perform the assessment bilaterally.
Participant functional performance | Change in functional performance over the course of active treatment.
  Subject's performance on the BBVR system will be recorded to gauge participant improvement on the BBVR system.
Participant symptoms | Change in symptom reporting from baseline to of the wait-list (for the wait-list control group only), midpoint (3 weeks) of active therapy, and end point (6 weeks) of active treatment.
  Post-Traumatic Stress Disorder (PTSD). The PTSD Checklist, Civilian Version (PCL-C) is a self-report questionnaire on the presence and severity of PTSD symptoms.
Participant symptoms | Change in symptom reporting from baseline to of the wait-list (for the wait-list control group only), midpoint (3 weeks) of active therapy, and end point (6 weeks) of active treatment.
  Neurobehavior Symptom Inventory. The Neurobehavioral Symptom Inventory (NSI) is routinely used as a standard assessment tool to gauge post-concussive symptoms of TBI.
Participant symptoms | Change in symptom reporting from baseline to of the wait-list (for the wait-list control group only), midpoint (3 weeks) of active therapy, and end point (6 weeks) of active treatment.
  Mood. Quick Inventory of Depressive Symptomatology, Self-Report (QIDS-SR) is a shortened version of the Inventory of Depressive Symptomatology, Self-report (IDS-SR) that covers just items that assess Diagnostics and Statistics Manual (DSM)-IV criterion diagnostic symptoms for depression.
Reliability of the BBVR technology when deployed in a clinical setting | Throughout the duration of the study - expected to last one year.
  Recording of BBVR Performance. A log of system reliability will be kept to determine mean time between failure and type of malfunction. To monitor computer usage, type of games played, and progress, each session will generate a paper-printed and a digital report.

CONTACTS AND LOCATIONS:
Overall Officials: Paul F Pasquina, MD, Principal Investigator — Walter Reed National Military Medical Center
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burdea G, Polistico K, Krishnamoorthy A, House G, Rethage D, Hundal J, Damiani F, Pollack S. Feasibility study of the BrightBrainer integrative cognitive rehabilitation system for elderly with dementia. Disabil Rehabil Assist Technol. 2015;10(5):421-32. doi: 10.3109/17483107.2014.900575. Epub 2014 Mar 29. PMID 24679074